CLINICAL TRIAL: NCT04458740
Title: The Life and Care of Colorectal Cancer Patients After 65 Years and Their Family
Acronym: MACHROAPIK65
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MACHROAPICANCERPLUS65
Record Dates: First submitted 2018-11-07; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Patients with a diagnosis of colorectal cancer after 65 years.
  Interventions: Other: biographical interviews
- The spouse and /or children and /or parents: The spouse and /or children and /or parents of a patient 's diagnosis of colorectal cancer before 65 years.
  Interventions: Other: biographical interviews

INTERVENTIONS:
Other: biographical interviews — A sociologist trained in the sociology of cancer, to enable participants to talk about their experiences and clearly distinguish the experiences of each individual

SUMMARY:
Given a context where patients autonomy respect is important, it is necessary to pay a sustained attention to the patients care and life experiences, as well as the families and relatives of patients with colorectal cancer or patients in remission of colorectal cancer. Thanks to families and relatives data, it will allow to improve the analyses carried out by the "Societal Cancer Observatory" in 2016.

ELIGIBILITY:
Inclusion Criteria:

The patients will be:

* over the age of 65 and under 80
* with a colorectal cancer operated between 65 and 80 years with a documented histological diagnosis, dating from 2 to 5 years.
* be able to provide informed consent and appoint a caregiver who would be willing to participate in the study.

The spouse and / or children and / or parents will be eligible:

if he is at least 18 years old, if he can be considered a caregiver of the index patient for whom a diagnosis of CRC has been made.

Exclusion Criteria:

* Patients with a diagnosis of colorectal cancer before the age of 65 or after the age of 80 from 2 to 5 years old.

Near a deceased patient or under 18 years old.

Ages: 65 Years to 80 Years | Sex: All
Age Groups: Older Adult
Study Population: Surviving patients between 65 and 80 years and diagnosed with invasive CRC, infiltrating adenocarcinoma of the colon or rectum irrespective of the stage before 65 years old will be selected in the Poitou-Charentes cancer registry 2 to 5 years after announcement of the diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-05-17 (Actual); Study Completion 2019-05-17 (Actual)

PRIMARY OUTCOMES:
Assess the interaction between the care path (surgery, chemotherapy, radiotherapy) and the life course in patients after 65 years old with colorectal cancer | 2 hours
  semi-structured patients interview
Assess how the patients and their family members face the disease | 1 hour
  semi-structured patients interview

CONTACTS AND LOCATIONS:
Locations (1):
- Registre du Cancer, Poitiers, France

IPD SHARING:
Plan to Share IPD: No